CLINICAL TRIAL: NCT06481579
Title: A Phase 2, Randomized, Modified Double-Blind, Active Controlled Study to Characterize the Safety and Immunogenicity of IVX-A12 in Adults 60 Years of Age and Older
Brief Title: A Study of IVX-A12 in Adults Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icosavax, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ICVX-12-202
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
Keywords: Respiratory syncytial virus (RSV); Human metapneumovirus (hMPV)
MeSH Terms: interventions — arexvy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVX-A12 Vaccine (Experimental): Participants will receive a single dose of IVX-A12, 300 micrograms (mcg), intramuscular (IM) injection on Day 1.
  Interventions: Biological: IVX-A12
- Licensed RSV Vaccine (Active Comparator): Participants will receive a single dose of licensed RSV vaccine (AREXVY) IM injection on Day 1.
  Interventions: Biological: Licensed RSV Vaccine

INTERVENTIONS:
Biological: IVX-A12 — IVX-A12 IM injection.
  Arms: IVX-A12 Vaccine
Biological: Licensed RSV Vaccine — Licensed RSV Vaccine (AREXVY) IM injection.
  Other Names: AREXVY
  Arms: Licensed RSV Vaccine

SUMMARY:
The primary purpose of this study is to assess the immunogenicity and safety of IVX-A12 in adults 60 years of age and older.

DETAILED DESCRIPTION:
This is a randomized, modified double-blind, active controlled study to characterize the immunogenicity and safety of IVX-A12.

Approximately 140 participants will be randomized in a 1:1 ratio to receive IVX-A12 (approximately 70) or licensed respiratory syncytial virus (RSV) vaccine (AREXVY) (approximately 70).

The study is planned to be conducted at approximately 5 sites in the United States. The duration of each participant's involvement in the study will be approximately 6 months following administration of study vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Adults >=60 years of age at the time of signing informed consent.
2. Participants who are medically stable according to the judgment of the Investigator.
3. Able to understand and comply with study requirements/procedures based on the assessment of the Investigator.
4. Capable of giving signed informed consent.

Exclusion Criteria:

1. Acute (time-limited) or febrile (temperature >=38.0 °C [100.4 ºF]) illness/infection within 3 days of planned dosing.
2. History of a clinically significant bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
3. History of hypersensitivity to any component of the study vaccination.
4. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis).
5. Known or suspected congenital or acquired immunodeficiency.
6. Known or suspected autoimmune condition as determined by history and/or physical examination.
7. History of Guillain-Barré syndrome or any other demyelinating condition.
8. History of malignancy other than treated non-melanoma skin cancers or locally-treated cervical cancer in previous 5 years.
9. Any condition that may significantly increase the risk to the participant because of participation in the study, impact the participant's ability to participate in the study, or impair the interpretation of the study data.
10. Receipt of any licensed or investigational RSV and/or Human metapneumovirus (hMPV) vaccine any time prior to administration of study intervention.
11. Receipt of any licensed vaccine (other than licensed influenza or COVID-19 vaccines) within 28 days prior to or expected receipt within 28 days after administration of study intervention. Licensed influenza or COVID-19 vaccines are permitted beginning greater than (>)14 days prior to and >14 days after administration of study intervention.
12. Receipt of immunoglobulin or blood products within 3 months prior to administration of study intervention or expected receipt during the study.
13. Receipt of immune-modifying drugs or immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy within 6 months prior to enrollment (or expected receipt during study), or long-term systemic corticosteroid therapy (prednisolone or equivalent at a dose of >=20 mg daily or every other day for more than 2 consecutive weeks) within 6 months prior to study intervention or anticipated receipt during study.
14. Participation in another study or receiving interventional study investigational medicinal product (IMP), in the preceding 28 days or expected receipt of another study intervention (or participation in another study) during the period of study follow-up.
15. Employees of the Sponsor involved in planning, executing, supervising, or reviewing the IVX-A12 program, clinical study site staff, or any other individuals involved with the conduct of the study, or immediate family members of such individuals.
16. Alcohol or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.
17. Deprived of freedom by an administrative or court order, or in emergency setting, or hospitalized involuntarily.
18. Judgment by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Icosavax Investigational Site US022, Anaheim, California
  - Icosavax Investigational Site US021, Rolling Hills Estates, California
  - Icosavax Investigational Site US002, Hollywood, Florida
  - Icosavax Investigational Site US011, Lenexa, Kansas
  - Icosavax Investigational Site US016, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 5 investigative sites in the United States.
Pre-assignment Details: A total 143 participants were enrolled and randomized to receive vaccinations in this study.
Groups:
- IVX-A12: Participants received a single dose of 300 micrograms (mcg) IVX-A12, intramuscular (IM) injection on Day 1.
- AREXVY: Participants received a single dose of 120 mcg AREXVY, IM injection on Day 1.
Period: Overall Study
Arm/Group | IVX-A12 | AREXVY
Started | 71 | 72
Completed | 66 | 71
Not Completed | 5 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety analysis set (SAF) included all randomized participants who received one dose of study intervention, irrespective of their protocol adherence and continued participation in the study.
Groups:
- IVX-A12: Participants received a single dose of 300 mcg IVX-A12, IM injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | IVX-A12 | AREXVY | Total
Number analyzed (Participants) | 71 | 72 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (5.9) | 66.6 (5.6) | 66.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 35 | 34 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 14 | 27
  Not Hispanic or Latino | 58 | 57 | 115
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 14 | 33
  White | 49 | 56 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Model-adjusted Geometric Mean Concentration (GMC) for RSV/A Neutralizing Antibodies (NAb)
Description: Model-adjusted GMCs and 95% CIs were derived using an ANCOVA model for log2 nAb responses at Day 29 with independent variables of study intervention, log2 baseline response, and age group. Measured values were calculated as the anti-logarithm transformation of the least square means and 95% CIs from the model.
Time Frame: At Day 29
Population: Immunogenicity analysis set (IAS) included all participants in the SAF who had no eligibility-related protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: internation unit per milliliter (IU/mL)
Arm/Group | IVX-A12 | AREXVY
Number analyzed (Participants) | 66 | 67
internation unit per milliliter (IU/mL) | 5910.4 [4210.4 to 8296.8] | 10500.4 [7565.2 to 14574.3]

2. Primary Outcome: Geometric Mean Fold Rise (GMFR) in RSV/A NAb Concentrations
Description: The GMFR was calculated as the anti-logarithm of Σ(log2 transformed (post-baseline response/baseline response)/n), where n is the number of participants with non-missing response information at baseline and at the post-baseline timepoint.
Time Frame: From baseline up to Day 29
Population: IAS included all participants in the SAF who had no eligibility-related protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | IVX-A12 | AREXVY
Number analyzed (Participants) | 66 | 67
fold rise | 3.4 [2.7 to 4.3] | 6.5 [5.0 to 8.5]

3. Primary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AEs)
Description: Immediate AEs were defined as having an onset time within 30 minutes after study vaccination.
Time Frame: Within the 30 minutes after vaccination on Day 1
Population: The SAF included all randomized participants who received one dose of study intervention, irrespective of their protocol adherence and continued participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | IVX-A12 | AREXVY
Number analyzed (Participants) | 71 | 72
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Injection Site and Systemic Solicited Adverse Reactions (ARs)
Description: The injection site solicited ARs included predefined injection site pain, injection site erythema/redness, and injection site swelling. The systemic solicited ARs included predefined fever, chills, headache, myalgia (muscle aches and pains), and fatigue (physical or mental tiredness).
Time Frame: Day 1 through Day 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | IVX-A12 | AREXVY
Number analyzed (Participants) | 71 | 72
Participants
  Solicited injection site AR | 14 | 31
  Solicited systemic AR | 19 | 17

5. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: The unsolicited AEs were any AE other than predefined solicited AEs.
Time Frame: Day 1 through Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | IVX-A12 | AREXVY
Number analyzed (Participants) | 71 | 72
Participants | 5 | 11

6. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Medically-attended Adverse Events (MAAEs), and Adverse Events of Special Interests (AESIs)
Description: A SAE defined as an AE that occurred during any phase of study and met one or more of following criteria: resulted in death; was immediately life-threatening; required in-patient hospitalization or led to prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; was a congenital anomaly or birth defect; or was considered an important medical event that might have jeopardized the participant or required medical intervention to prevent one of aforementioned outcomes. MAAEs defined as AEs leading to medically-attended visits that were not routine visits for physical examination or vaccination, such as an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. An AESI was an event of scientific and medical interest, specific to further understanding of safety profile of investigational vaccine and required close monitoring and rapid communication by Investigators to the Sponsor.
Time Frame: Day 1 through Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | IVX-A12 | AREXVY
Number analyzed (Participants) | 71 | 72
Participants
  SAEs | 2 | 1
  MAAEs | 1 | 9
  AESIs | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through Day 181
Arm/Group | IVX-A12 | AREXVY
All-Cause Mortality (participants affected / at risk) | 1/71 | 0/72
Serious Adverse Events (participants affected / at risk) | 2/71 | 1/72
Other Adverse Events (participants affected / at risk) | 6/71 | 15/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVX-A12 (N=71) | AREXVY (N=72)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVX-A12 (N=71) | AREXVY (N=72)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 1 (1) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT06481579/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT06481579/SAP_001.pdf